CLINICAL TRIAL: NCT07168031
Title: Neural and Age-Related Effects of Transcranial Direct Current Stimulation of the Left dlPFC During Information Processing
Brief Title: tDCS of the Left dlPFC: Effects on Information Processing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 50012
Record Dates: First submitted 2025-08-28; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Non-invasive brain stimulation; tDCS; fMRI; dlPFC; Hippocampus; Ageing; Neuroimaging

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded to the stimulation condition. Both active and sham tDCS procedures involve identical electrode placement and an initial ramp-up of current to produce similar sensations. In the sham condition, the current is turned off after the ramp-up period, preventing ongoing stimulation while maintaining the same setup and experience for participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS of the Left dlPFC (Experimental): Participants receive active anodal tDCS over the left dorsolateral prefrontal cortex during an information processing task for 22 minutes at 1 mA, with a gradual ramp-up and ramp-down of 30 seconds at the beginning and end of the stimulation.
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS of the Left dlPFC (Sham Comparator): Participants receive sham tDCS with the same setup and initial ramp-up of current to mimic the sensation of active stimulation. The current is turned off after the ramp-up period, and no further stimulation is delivered during the task.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — High definition tDCS will be applied, using a Soterix Medical device and 4x1 ring electrodes. A centre ring electrode overlying the target cortical region (left dlPFC at position F3 according to the 10-20 system) will be surrounded by four return electrodes (position F1, FC3, F5, and AF3).
  Arms: Active tDCS of the Left dlPFC
Device: Sham Transcranial Direct Current Stimulation (tDCS) — The same setup and device as in the active tDCS group will be used, but in this case stimulation will be turned off after a ramp-up phase of 30 seconds. This mimics the same sensory feeling as active tDCS.
  Arms: Sham tDCS of the Left dlPFC

SUMMARY:
This study investigates how a non-invasive form of brain stimulation, called transcranial direct current stimulation (tDCS), affects brain activity and information processing in younger and older adults. The stimulation uses a very weak electrical current applied through electrodes placed on the scalp. This method is safe and widely used in research to study brain function.

Participants will complete computer-based tasks while receiving either active brain stimulation or a placebo (sham) stimulation. The task is designed to engage specific mental processes so that the investigators can study how the brain responds under different conditions. Brain activity will be measured using magnetic resonance imaging (MRI), both while participants perform the tasks and while they are resting.

The study will compare healthy younger (ages 20-40) and older (ages 60-80) adults to explore whether age influences how the brain responds to stimulation. By examining patterns of brain activation and connectivity, the investigators aim to better understand how tDCS can modulate cognitive processing across the adult lifespan.

The hypothesis is that applying tDCS to the left dorsolateral prefrontal cortex will change patterns of brain activity related to cognitive processing, and that these changes may differ between younger and older adults. This knowledge could help inform future research into brain stimulation techniques in different age groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy younger adults (ages 20-40) or healthy older adults (ages 60-80)
* Normal or corrected-to-normal vision and hearing
* Right-handed (for consistency in brain stimulation)
* Able to give written informed consent and comply with study procedures

Exclusion Criteria:

* History of neurological or psychiatric disorders
* Current use of medications that affect the central nervous system
* Metal implants, pacemakers, or other contraindications for MRI or tDCS
* History of seizures or epilepsy
* Pregnancy
* Participation in another brain stimulation study within the last 3 months
* Any condition judged by investigators to interfere with safe participation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Task Accuracy | During the intervention
  Accuracy in responses during an information processing task, measured as the proportion of correct responses.
Task-Related Brain Activation | During the intervention
  Changes in blood-oxygen-level-dependent (BOLD) signal during the information processing task, measured using fMRI.
Resting-State Functional Connectivity | Immediately before and after the intervention
  Changes in functional connectivity between brain regions before and after stimulation, measured using resting-state fMRI.

SECONDARY OUTCOMES:
Task Reaction Time | During the intervention
  Time in milliseconds between stimulus presentation and participant response during the information processing task.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Peter, Prof., Principal Investigator — UniversityClinics, University of Bern
Locations (1):
- University of Bern, Department of Old Age Psychiatry and Psychotherapy, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No